CLINICAL TRIAL: NCT06160362
Title: The Safety and Efficacy of Double-target CART-19 and 20 Cells in Relapse and Refractory Patients With CD19+/CD20+ Non-Hodgkin's Lymphoma (NHL)
Brief Title: The Safety and Efficacy of Double-target CART-19 and 20 Cells in Non-Hodgkin's Lymphoma (NHL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhihua Yao, PhD, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Th_C155
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: non-Hodgkin's lymphoma; CART
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- double-target CART-19 and 20 (Experimental): Patients will receive a pre-conditioning with cyclophosphamide and fludarabine before infusion of double-target CART-19 and 20 cells. The double-target CART-19 and 20 cells are to be administered on day0.
  Interventions: Biological: CART-19 and 20 cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: CART-19 and 20 cells — Double-target CART-19 and 20 cells will be administered on day0 after completion of the chemotherapy.
Drug: Cyclophosphamide — patients will receive a standard pre-conditioning regime with cyclophosphamide 500mg/m2/day IV for 2 days(Day-3 to day-2).
Drug: Fludarabine — Fludarabine 25mg/m2/day IV for 3 days (Day-4 to day-2).

SUMMARY:
This is a study for patients who have been previously treated for NHL. The purpose of this study is to determine the safety and feasibility of double-target CART-19 and 20 cells to the patients with relapsed and refractory CD19+/CD20+ NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old (including 18 and 75)
2. Diagnosed as R/R NHL
3. CD19/CD20 positive confirmed by cell flow cytometry or immunohistochemistry
4. Having at least one measurable lesions
5. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2
6. Life expectancy no less than 3 months
7. enough main organ function
8. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and 12 months after this study
9. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 12 months
2. Active GVHD
3. History of severe pulmonary dysfunction
4. Active malignant tumor need be treated at the same time
5. Uncontrolled active acute/chronic infection
6. Severe autoimmune diseases or congenital immunodeficiency
7. Untreated active hepatitis
8. HIV-positive, AIDS patients and syphilis infection
9. History of severe allergies to biological products
10. Patients with a history of mental illness
11. Pregnant or lactating women; (female participants of reproductive potential must have a negative serum or urine pregnancy test)
12. Researchers think of that does not fit to participate in the study, or other cases that affect the clinical trial results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
safety as assessed by the occurrence of study related adverse events | from the date of recieving intravenous CART cells up to one month
  monitor the occurrence of study related adverse events

SECONDARY OUTCOMES:
objective response rate | 28 days and 3 months after recieving intravenous CART cells
  the proportion of patients benefit from the therapy
peripheral blood CART cell copy number | from the date of recieving intravenous CART cells up to one month
  The highest concentration of CART cells in peripheral blood, the time to reach the highest concentration, and the area under the curve at 28 days after recieving intravenous CART cells

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Yao, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China